CLINICAL TRIAL: NCT03137186
Title: Mansmed Trial : Repurposing Metformin as Anticancer Drug, RCT in Advanced Prostate Cancer
Brief Title: Repurposing Metformin as Anticancer Drug: in Advanced Prostate Cancer
Acronym: Mansmed
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Reham Algahndour, Assistant lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mansmed trial I
Record Dates: First submitted 2017-04-09; First posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: Metformin, prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Investigational arm (Active Comparator): Metformin will be added to standard of care
  Interventions: Drug: Metformin
- Control arm (No Intervention): Patients will treated according to Standard of care only

INTERVENTIONS:
Drug: Metformin — Metformin will be added as a daily treatment to the standard treatment in both neoadjuvant and adjuvant settings of locally advanced cases and lifelong to metastatic cases. The starting daily dose of metformin is 850mg Once daily, to be increased to 850 mg if tolerated
  Other Names: Cidophage
  Arms: Investigational arm

SUMMARY:
This study evaluate the addition of metformin to standard of care in locally advanced and metastatic prostate cancer, half the patient will receive metformin in combination with standard treatment, and the other half will receive the standard of care only

DETAILED DESCRIPTION:
Advanced-stage PCa is usually treated with androgen-deprivation therapy (ADT). Most patients with metastatic disease who were managed with ADT eventually progress to castration-resistant prostate cancer (CRPC) and die of the disease. CRPC can be treated with docetaxel, abiraterone plus prednisone, enzalutamide, and cabazitaxel, which provide limited survival benefits. Thus, there is still a need to improve the therapeutic options available for advanced-stage prostate cancer patients. Targeting therapy-resistant cancer stem cells (CSCs )in prostate cancer provides a unique opportunity for novel therapeutic interventions.

Metformin, a common well-tolerated oral biguanide prescribed for type II diabetes, could be used to sensitize prostate CSCs to current conventional anticancer therapies and improve the efficacy of treatment. Some studies reported that Metformin could enhance the effectiveness of ADT. Metformin augmented the antiproliferative and apoptotic effects of ADT in prostate cancer. The combination of these two drugs significantly reduces prostate cancer cell growth compared to monotherapy with either drug. Also, metformin might reduce the development of CRPC.

Many studies showed that obesity and DM were linked to aggressive prostate cancer phenotype, including biochemical failure after radical prostatectomy and external beam radiotherapy with higher incidence of complications of ADT. Interestingly, metformin reduces the incidence of diabetes and the adverse metabolic effects of ADT, including hyperinsulinaemia and dyslipidaemia, and decreases myocardial infarction risk and prolongs survival in diabetic patients.

To the best of our knowledge, after extensive computer research, there is no published results from prospective randomized trials evaluating role of metformin among men with high risk locally advanced or metastatic prostate cancer patients who will start treatment with ADT.

ELIGIBILITY:
Inclusion Criteria:

1. High-risk newly diagnosed non-metastatic node-negative disease at least two of:

   * Stage T3/4, PSA≥40ng/ml or Gleason sum score 8-10
   * Intention to treat with radical radiotherapy (unless there is a contraindication)
2. OR newly diagnosed metastatic or node-positive disease at least one of:

   * Stage T any N+ M0
   * Stage T any Nany M+
3. OR previously treated with radical surgery and/or radiotherapy, now relapsing

   At least one of:

   (-PSA ≥4ng/ml and rising with doubling time less than 6 months,N+, M+)
4. And for all patients

   * Age > 18 years
   * Histologically confirmed prostate adenocarcinoma
   * Intention to treat with long-term androgen deprivation therapy
   * Fit for all protocol treatment and follow-up, ECOG performance status 0-2
   * Diabetic and non-diabetic patients
   * Patients with adequate organ function(AST - ALAT ≤ 2.5x ULN,Bilirubin ≤ 1.5 x ULN)

Exclusion Criteria:

1. Age < 18 years
2. Excessive alcohol intake, acute or chronic
3. Patients already treated with Metformin or an analoge
4. Known hypersensitivity or allergy to Metformin or any of the excipients.
5. Patients with a history of lactic acidosis
6. Patient treated for a cancer other than prostate cancer, with the exception of basal cell carcinoma
7. Acute or chronic metabolic acidosis.
8. Patients suffering from severe dehydration.
9. Patients with chronic heart failure.
10. Patients with hepatic impairment.
11. Patients with severe renal disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
duration in months from beginning of treatment till development of CRPC | 2 years
  time till development of CRPC [Castrate resistant prostate cancer], is defined by disease progression despite androgen depletion therapy (ADT) and may present as either a continuous rise in serum prostate-specific antigen (PSA) levels, the progression of pre-existing disease, and/or the appearance of new metastases.

SECONDARY OUTCOMES:
CRPC free survival | 4 years
  Number of survivors without CRPC at 4 years
Overall patients' survival | 4 years
  Number of overall survivors at 4 years regardless occurrence of CRPC or not

CONTACTS AND LOCATIONS:
Overall Officials: Reham Alghandour, Principal Investigator — Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Colquhoun AJ, Venier NA, Vandersluis AD, Besla R, Sugar LM, Kiss A, Fleshner NE, Pollak M, Klotz LH, Venkateswaran V. Metformin enhances the antiproliferative and apoptotic effect of bicalutamide in prostate cancer. Prostate Cancer Prostatic Dis. 2012 Dec;15(4):346-52. doi: 10.1038/pcan.2012.16. Epub 2012 May 22. PMID 22614062
- [Result] Dowling RJ, Goodwin PJ, Stambolic V. Understanding the benefit of metformin use in cancer treatment. BMC Med. 2011 Apr 6;9:33. doi: 10.1186/1741-7015-9-33. PMID 21470407
- [Result] Eriksson A, Attvall S, Bonnier M, Eriksson JW, Rosander B, Karlsson FA. Short-term effects of metformin in type 2 diabetes. Diabetes Obes Metab. 2007 Jul;9(4):483-9. doi: 10.1111/j.1463-1326.2006.00624.x. PMID 17587390
- [Result] Hamilton RJ. Metformin for castrate-resistant prostate cancer: learning more about an old dog's new tricks. Eur Urol. 2014 Sep;66(3):475-7; discussion 477-8. doi: 10.1016/j.eururo.2014.01.013. Epub 2014 Jan 23. No abstract available. PMID 24472709
- [Result] Hankinson SJ, Fam M, Patel NN. A review for clinicians: Prostate cancer and the antineoplastic properties of metformin. Urol Oncol. 2017 Jan;35(1):21-29. doi: 10.1016/j.urolonc.2016.10.009. Epub 2016 Nov 9. PMID 27836248
- [Result] Mayer MJ, Klotz LH, Venkateswaran V. Metformin and prostate cancer stem cells: a novel therapeutic target. Prostate Cancer Prostatic Dis. 2015 Dec;18(4):303-9. doi: 10.1038/pcan.2015.35. Epub 2015 Jul 28. PMID 26215782
- [Result] Ranasinghe WK, Sengupta S, Williams S, Chang M, Shulkes A, Bolton DM, Baldwin G, Patel O. The effects of nonspecific HIF1alpha inhibitors on development of castrate resistance and metastases in prostate cancer. Cancer Med. 2014 Apr;3(2):245-51. doi: 10.1002/cam4.189. Epub 2014 Jan 27. PMID 24464861
- [Result] Rothermundt C, Hayoz S, Templeton AJ, Winterhalder R, Strebel RT, Bartschi D, Pollak M, Lui L, Endt K, Schiess R, Ruschoff JH, Cathomas R, Gillessen S. Metformin in chemotherapy-naive castration-resistant prostate cancer: a multicenter phase 2 trial (SAKK 08/09). Eur Urol. 2014 Sep;66(3):468-74. doi: 10.1016/j.eururo.2013.12.057. Epub 2014 Jan 4. PMID 24412228
- [Result] Saylor PJ, Smith MR. Metabolic complications of androgen deprivation therapy for prostate cancer. J Urol. 2009 May;181(5):1998-2006; discussion 2007-8. doi: 10.1016/j.juro.2009.01.047. Epub 2009 Mar 14. PMID 19286225
- [Result] Song CW, Lee H, Dings RP, Williams B, Powers J, Santos TD, Choi BH, Park HJ. Metformin kills and radiosensitizes cancer cells and preferentially kills cancer stem cells. Sci Rep. 2012;2:362. doi: 10.1038/srep00362. Epub 2012 Apr 12. PMID 22500211
- [Result] Spratt DE, Zhang Z, Zelefsky MJ. Reply to Leah Bensimon, Samy Suissa, and Laurent Azoulay's letter to the editor re: Daniel E. Spratt, Chi Zhang, Zachary S. Zumsteg, Xin Pei, Zhigang Zhang, Michael J. Zelefsky. metformin and prostate cancer: reduced development of castration-resistant disease and prostate cancer mortality. Eur Urol 2013;63:709-16. Eur Urol. 2013 Aug;64(2):e29-30. doi: 10.1016/j.eururo.2013.04.015. Epub 2013 Apr 19. No abstract available. PMID 23619389
- [Result] Heidenreich A, Bastian PJ, Bellmunt J, Bolla M, Joniau S, van der Kwast T, Mason M, Matveev V, Wiegel T, Zattoni F, Mottet N; European Association of Urology. EAU guidelines on prostate cancer. Part II: Treatment of advanced, relapsing, and castration-resistant prostate cancer. Eur Urol. 2014 Feb;65(2):467-79. doi: 10.1016/j.eururo.2013.11.002. Epub 2013 Nov 12. PMID 24321502